CLINICAL TRIAL: NCT06258512
Title: Impact of an Intervention with a Narrative Approach in Overusers in Primary Health Care: a Controlled and Randomized Trial
Brief Title: Impact of an Intervention with a Narrative Approach in Overusers: a Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Catalan Institute of Health (Other Government)
Responsible Party: Principal Investigator, Valentin Calvo Rojas, Principal Investigator, Catalan Institute of Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CatalanIH
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Overuse Syndrome
Keywords: Healthcare utilisation; Psychosocial determinants of health; Primary care; Affective social support; Frequent attenders
MeSH Terms: conditions — Cumulative Trauma Disorders | interventions — Methods; Narrative Therapy

STUDY DESIGN:
Intervention Model Description: The interventions of the health social workers rely on listening in the clinical interview, They give space to the patient's subjective complaint, they locate the understanding of the discomfort and the symbolic meaning of the symptoms. The difficulties are focused as elements of the relationship between the professional and the user and does not refer to pharmacological treatments. Since social work identifies discomfort psychosocial as an object of study, we would like to demonstrate that, establishing locally an intervention with a narrative approach implemented in the area of primary health care with the aim of improving the perception of emotional support of users with excessive use of self-initiated consultation, we can reduce the use of medical consultations, and, most importantly, the suffering and discontent of said users who do not find an answer appropriate to your discomforts.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention with narrative approach + standard care (Experimental): Intervention with a narrative approach. The objectives will be:
  1. Know significant moments in the personal history of the participant and her family according to her life cycle. as well as structural elements.
  2. Know information regarding symptoms of non-organic origin, pain crises, personal and family resources for their management.
  3. Implement a narrative technique as an alternative for the management of symptoms of non-organic origin, including the following strategies: the participant will be able to tell and retell their story, recognize situations or moments that exacerbate the pain, feel the pain and name it, externalization of the pain. problem, the problem is the problem, absolving oneself from traumatic life experiences, constructing meaning to one's dominant stories through the organization of the experience, to obtain a new meaning of what was experienced through the story, construction of alternative stories.
  Interventions: Other: Intervention with a narrative approach.
- control with standard care (No Intervention): Participants randomly assigned to the control group will receive usual care from their primary care professionals.

INTERVENTIONS:
Other: Intervention with a narrative approach. — Health social workers will carry out a intervention with a narrative approach, through its training profile based on transversal skills, which will consist of 10 sessions carried out over five months. The interval between sessions will be of two weeks with a specific duration of fifty minutes per session. This type of intervention, with the objective of reorienting and redefining the demand or the initial problems that motivated the consultation, gives space to the patient's subjective complaint, as well as to locate the understanding of the discomfort and the symbolic meaning of the symptoms.
  That is, recognizing the physical symptoms while listening to stories of chaos to legitimize both the user and his symptoms, an encounter that allows return the user to its context without feeling rejected or judged by the health system.
  Other Names: Narrative therapy
  Arms: Intervention with narrative approach + standard care

SUMMARY:
The goal of this clinical trial is to compare an intervention with a narrative therapy-based approach with standard care in overusers in general practice . The main question it aims to answer are:

• An intervention with an approach based on narrative therapy can improve the perception of emotional support, and reduce the probability of suffering from anxiety and/or depression, the number of consultations, and the number of medications in primary care overusers.

Participants will 10 individual sessions carried out over five months. The interval between sessions will be two weeks with a specific duration of fifty minutes per session..

If there is a comparison group: Researchers will compare two groups of overusers to see if reduces the number of visits to the primary care doctor.

DETAILED DESCRIPTION:
Background: The best treatment for the excessive use of the consultation is currently being discussed.

Hypothesis: An intervention with an approach based on narrative therapy, compared to standard care, leads to reducing psychosocial distress and reducing the number of consultations with the family doctor.

Objective: To evaluate the effectiveness of an intervention based on co-constructing a new narrative of symptoms of non-organic origin compared to usual clinical care, with respect to affective social support, the probability of suffering from anxiety and/or depression, and the use of the medical consultation.

Methodology: Pragmatic, controlled and randomized, non-masked clinical trial. Study subjects: 264 users (132 in each group, intervention and control) with excessive use of the consultation (95th percentile of the distribution of appointment-type and/or urgent visits to the medicine service). Intervention will be compared with narrative approach + standard care / standard care.

Determinations: Symptoms of anxiety and depression, social support, number of consultations, age, sex, marital status, educational level, income level, employment status.

Statistical analysis: In order to determine the discriminant capacity of the variables associated with the intervention, we will build a multiple regression model in which we will include those that were statistically significant in the bivariate analysis and those that are relevant according to the bibliography.

Expected results: The results will provide evidence on the effectiveness of said intervention.

Application and Relevance: This type of intervention would most likely reduce the pressure on medical-health professionals.

ELIGIBILITY:
Inclusion Criteria:

* Users in the 95th percentile in the distribution of consultations face-to-face, patient self-initiated consultations with PHC services within the period of 1 year.

Exclusion Criteria:

* Drug abuse or dependence, except for nicotine and tetrahydrocannabinol.
* Comorbidity with DSM-IV-TR (American Psychiatric Association, 2000) severe mental disorders.
* Comorbidity with ICD-10 (World Health Organization, 2008) severe cognitive disorders or sensory disabilities.
* Major locomotor mobility limitations or terminal illness

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2023-10-18 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in affective social support at 1 month, 6 months, and 18 months | Before randomization and at the end of treatment at 1 month, six months and 18 months
  - Health-related social support: Affective social support: between 5-14 poor social support / between 15 and 25 good social support. Confidential social support: between 6-17 no confidential social support / between 18 and 30 good social support. Total social support: between 11-32 no social support / between 33-55 social support It is a variable that values people's perception, from a person-centered approach to care: For its measurement we will use the DUKE-UNC functional social support scale. This is a questionnaire self-assessment consisting of 11 items that evaluates perceived social support using a five-point Likert scale. This scale provides three indicators: Affective social support with a range between 25 and 5, being the point of cut of 15; Confidential social support with a range between 30 and 6 points, being cut-off point of 18 and total social support with a range between 55 and 11 points, the cut-off point being 33. If the final score is below 33, the considers absence

SECONDARY OUTCOMES:
Change from baseline in probability of having an anxiety or depressive at 1 month, 6 months, and 18 months | Before randomization and at the end of treatment at 1 month, six months and 18 months
  Goldberg Anxiety-Depression Scale. This is an 18-item self-report symptom inventory with a yes/no response format (Yes = 1, No = 0). The scores are based on responses to nine anxiety and nine depression items, asking how respondents have felt in the past month. The cut-off points of the Spanish version are ≥4 for anxiety and ≥2 for depression; higher scores are indicative of a high probability of having an anxiety or depressive disorder. This scale orients the diagnosis towards anxiety or depression, or both in mixed cases, and discriminates between the two entities while measuring their respective intensities,
Change from baseline in variables related to drug exposure at 1 month, 6 months, and 18 months | Before randomization and at the end of treatment at 1 month, six months and 18 months
  Drug exposure is analyzed through the primary care medical history prescription database. This database contains all medications dispensed by pharmacies. Medicines are classified according to the anatomical-therapeutic classification system: • Number of medications. We classified patients into five categories according to the number of different pharmaceutical specialties that the patient has been prescribed: 0; 1; 2 to 4; 5 to 9; 10 or more. • Prescription of anxiolytic and antidepressant drugs: the following therapeutic groups of interest are identified according to ATC classification: o Anxiolytics and hypnotics: N05BA Benzodiazepine derivatives; N05CD Benzodiazepine derivatives; N05CF Benzodiazepine-related drugs; N05CH Melatonin receptor agonists; N03AE01 Clonazepam (clonazepam is included given its high use as an anxiolytic and hypnotic agent) o Antidepressants: N06AB Selective serotonin reuptake inhibitors; N06AX Other antidepressants
Number of visits patient self-initiated consultations with PHC services, and totals, per year | Before randomization and at the end of treatment at 1 month, six months and 18 months
  They will be extracted from the electronic medical records

OTHER OUTCOMES:
Sociodemographic data | Before randomization
  We collected the following variables: Age, gender, civil status, educational level, monthly income, employment status, family life cycle and family structure. Employment status was categorised as being active in the workforce with paid work (employee or employer) or inactive/unemployed. Family life cycle was categorised as Stage I (couples with no children); Stage II (couples with children); Stage III (middle-aged parents: stage begins with empty nest) and Stage IV (aging family members: stage begins with spouses' retirement and ends at their deaths). Family structure was categorised as living alone (without close relatives but may share housing with other relations), nuclear family (including single-parent families) and extended family (enlarged nuclear family, including relatives).
Clinical variables | Before randomization
  The following symptoms and functional syndromes of interest are identified, which will be extracted from the record of the list of active problems in the computerized medical history: Musculoskeletal pain; Tiredness/asthenia; Headache/migraine/migraine; Dizziness/vertigo; Sleep disturbance/insomnia/difficulty sleeping; Palpitations/tachycardia; Fibromyalgia; Decreased appetite; Dyspnea/difficulty breathing; Irritable Colon; Abdominal pain; Chronic fatigue; Nausea/vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre d'Atenció Primària Montnegre, Institut Català de la Salut, Barcelona, Catalonia, Spain, Barcelona, Catalonia, Spain

IPD SHARING:
Plan to Share IPD: No